CLINICAL TRIAL: NCT05434338
Title: Study of the Dynamics of Human Papillomavirus (HPV) Clearance in Post-treatment of High-grade Intraepithelial Lesions (HGIL).
Brief Title: Papillomavirus Post-THErapeutique
Acronym: PAPOTHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220619
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: High Grade Intraepithelial
Keywords: conization; high-grade intraepithelial lesion (HGILs); post-therapy HPV clearance; HPV test; disappearance kinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Major women with HPV-related high-grade intraepithelial lesions (Other)
  Interventions: Diagnostic Test: HPV detection test

INTERVENTIONS:
Diagnostic Test: HPV detection test — Samples taken from the squamocolumnar junction using swabs (UTM Copan)
  Other Names: PCR HPV test [AnyplexTM HPV28 Detection (Seegene®)] : swab UTM Copan

SUMMARY:
In recent years, studies have multiplied to demonstrate the value of performing an HPV test compared to a cervical smear test (CSP) in cervical cancer screening but also in the follow-up of surgical removal of high-grade intraepithelial lesions (HGILs). Thus, since June 2019, the High Health Authority recommends performing HPV genome testing by PCR for primary cervical cancer screening. Since September 2019, the National Cancer Institute recommends an HPV test in the follow-up of HGILs 6 months after conization. However, this delay was determined thanks to the previous recommendations which advocated a cervical smear test 6 months after conization. Thus, the kinetics of HPV clearance in the immediate postoperative period and in the 6 months following surgical excision remain unknown to this day. A better knowledge of the clearance of HPV postoperatively would allow to adapt and simplify the follow-up of the patients and to personalize it according to the type of HPV.

DETAILED DESCRIPTION:
For research purposes, on the day of surgery, specimens at the squamocolumnar junction intraoperatively before and after surgical removal of the HGILs will be taken. Then at follow-up visits at M1 (care, +/-3 weeks), M3 (research, +/- 6 weeks), M6 (care, +/- 6 weeks), and M12 (care, +/- 6 weeks), two types of sampling will be performed :

* A self-sampling, performed by the patient at the vaginal level during the follow-up consultations (before the gynecological examination)
* After the speculum has been inserted, a swab sample will be taken by the doctor at the squamocolumnar junction. This procedure will be carried out before any other procedures expected as part of the treatment [colposcopy +/- biopsy(s)], All of these samples for HPV testing will be sent to the virology laboratory of the Pitié Salpêtrière Hospital, where they will be stored and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over 18 years old
* High-grade intraepithelial lesion (WHO classification)
* Intracervical neoplasms 2 and 3, Richart classification
* Collection of written, free and informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Immunocompromised patients (HIV infection, or iatrogenic)
* Patient with a history of treated HGIL
* Patient who does not understand French
* Patient unable to express consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the percentage of patients treated surgically for HGILs with a negative HPV PCR sample | immediate postoperative period
  The negativity rate will be described using a frequency, with a 95% confidence interval.

SECONDARY OUTCOMES:
determine if HPV PCR negativity in the immediate postoperative period is associated with persistence of negativity at 6 months. | immediate postoperative and at 6 months
  compare HPV PCR immediately postopertive and at 6 month
Describe postoperative HPV PCR kinetics according to HPV type. | at 1 month, 3 months , 6 months and 12 months
  Compare type of HPV determined on postoperative HPV PCRat 1 month, 3 months , 6 months and 12 months
Evaluate the association between the result of the HPV PCR in the immediate postoperative period and the rate of risk of relapse/persistence of LIEHGs in the year following the treatment. | immediate postoperative and at 12 months
  compare results of HPV PCR performed immediately postoperatively and at 12 months
Assess the association between the date of positivity of the HPV PCR and a risk of recurrence/persistence of high-grade dysplasia over the one-year follow-up period. | at 12 months
  calculation of the time between HPV PCR positivity at follow-up and development/persistence of high-grade dysplasia on biopsy over the one-year follow-up period
Evaluate the evolution of the negativity of the HPV tests at 0, 1, 3, 6 and 12 months in order to define an optimized follow-up. | immediately after surgery and at 1 month, 3 months , 6 months and 12 months
  comparison of the negativity of the HPV PCR performed immediately after surgery, at 1 month, 3 months , 6 months and 12 months
Compare the performance of the results of the PCR HPV Autotests and PCR HPV tests carried out by the practitioner. | at 1 month, 3 months , 6 months and 12 months
  comparison of patient self-test results at 1 month, 3 months , 6 months and 12 months prior to the consultation
Determination of the real risk of lesion persistence and consider de-escalation monitoring via the sorting of positive HPV-HR by a cytochemical study (p16 and Ki67). | at 12 months
  Number of participants with additional cytochemical study ( p16 and Ki67) in case of positive HPV tests with high risk HPV

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy Canlorbe, MD, PhD, Study Chair — APHP
Locations (1):
- Service : Chirurgie et oncologie gynécologique et mammaire, Hôpital Pitié Salpêtrière, Paris, France